CLINICAL TRIAL: NCT01566734
Title: Comparison of the Effect of Cefazolin and Normal Saline Irrigation With no Irrigation on the Incidence of Surgical Site Infections
Brief Title: Effect of Cefazolin and Normal Saline Irrigation on Surgical Site Infections (SSIs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hormozgan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mohammad E Shahrzad, MD, Mohammad Esmaeil Shahrzad, Hormozgan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: U1111-1128-4677
Record Dates: First submitted 2012-03-26; First posted 2012-03-29 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: Surgical Site Infections
Keywords: Surgical Wound Infection; cefazolin; Cesarean Section
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cefazolin; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cefazolin (Experimental): after the surgery and before closing up the patients, 2 grams of cefazolin in 5 cc of distilled water was used to irrigate the patients
  Interventions: Other: Cefazolin irrigation
- Normal Saline (Experimental): after the surgery and before closing up the patients, 150 cc of normal saline was used to irrigate the patients
  Interventions: Other: Normal Saline Irrigation
- Control (No Intervention)

INTERVENTIONS:
Other: Cefazolin irrigation — after the surgery and before closing up the patients, 2 grams of cefazolin in 5 cc of distilled water was used to irrigate the patients
  Other Names: cephazolin; cefazoline; Ancef; Cefacidal; Cefamezin; Cefrina; Elzogram; Faxilen; Gramaxin; Kefazol; Kefol; Kefzolan; Kezolin; Novaporin; Reflin; Zinol; Zolicef
  Arms: Cefazolin
Other: Normal Saline Irrigation — after the surgery and before closing up the patients, 150 cc of normal saline was used to irrigate the patients and in the last group
  Other Names: sodium chloride; saline solution
  Arms: Normal Saline

SUMMARY:
This study conducted to assess the effects of normal saline or cefazolin irrigation on the incidence of SSIs.

Hypothesis:

Normal saline or cefazolin irrigation decreases the incidence of SSIs.

DETAILED DESCRIPTION:
All pregnant women who underwent cesarean after 6 hours passed their rupture of membrane and attended to Shariati Hospital of Bandarabbass were eligible for our study.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* 6 hours passed their rupture of membrane
* needed to undergo cesarean

Exclusion Criteria:

* allergy to penicillin
* allergy to cefazolin
* history of immunosuppressive drug use
* gestational diabetes mellitus
* preeclampsia

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
SSI | one week after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Rahmani, MD, Study Director — Hormozgan University of Medical Sciences
Locations (1):
- Shariati Hospital, Bandar Abbas, Hormozgan, Iran